CLINICAL TRIAL: NCT06074770
Title: Study on Dietary Intake Levels of Iodine for 3-6 Years Old Pre-school Children
Status: Recruiting | Type: Observational
Sponsor: Chen Wen (Other)
Collaborators: Shandong Institute for Endemic Disease Control and Research (Unknown)
Responsible Party: Sponsor-Investigator, Chen Wen, associate professor, Tianjin Medical University
Organization: Tianjin Medical University (Other)
Other Study IDs: NSFC-8227121511
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Nutritional Requirements
Keywords: nutrient; dietary intake levels; pre-school children; iodine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 1. A 7-day iodine balance experiment was conducted in pre-school age children with insufficient iodine nutrition. Dietary intervention with different iodine intake, daily food and drinking iodine intake was accurately measured by double meal method, and 24-h urine and feces were collected for the measurement of iodine excretion
  2. The epidemiological survey of preschool children aged 3-6 years was carried out in high water iodine areas of Shandong Province, the iodine intake was accurately assessed through dietary survey and 24-h urine samples, and the thyroid volume, thyroglobulin and growth and development were measured to evaluate the effect of long-term high iodine exposure on preschool children
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — Natural exposure of iodine

SUMMARY:
Iodine as an essential trace element for human, both excessive and insufficient intake would be harmful for human health. As susceptible population, children will be more sensitive to adverse effects caused by inadequate intake of iodine since they are at the peak of growth and development. Meanwhile, there are few direct evidence to establish dietary intakes levels of iodine for 3-6 years old pre-school children.

DETAILED DESCRIPTION:
This study plan to conduct iodine balance experiment by providing devised diet consist of different iodine contents, in order to simulate iodine equilibrium of iodine deficiency to iodine excess in children and find the lowest iodine requirement of iodine for pre-school children, then aim to provide data to establish recommend nutrient intake of iodine for 3-6-year-old pre-school children. On the other hand, this study will make use of natural geographic environment with high water iodine in China. The investigators will conduct big-scale epidemiologic study in areas with high water iodine levels in Shandong and areas with adequate iodine in Tianjin, to enroll pre-school children with various iodine intake levels. The investigators will collect 24-hour urine samples as well as dietary records to evaluate iodine intake levels, and detect thyroid volume and thyroglobulin to evaluate the effects of various iodine intake on pre-school children, aiming to find the lowest safe intake level of iodine and then establish the tolerable upper intake level (UL) of iodine for 3-6-year-old pre-school children. This study aims to define the RNI and UL of iodine for 3-6-year-old pre-school children, to provide data for revision of Chinese dietary intake levels of iodine, and to guide children safe and scientifical iodine fortification.

ELIGIBILITY:
Inclusion Criteria:

* for children with mild malnutrition: hemoglobin <110g / L, or weight for age <P50 according to the Chinese 2009 child growth and development reference standard, or BMI z score <-1 according to the WHO Child Growth Assessment Software (version 3.2.2 ) ; have not been treated for thyroid disease; have not used amiodarone and other drugs (including iodine supplements) during the investigation; have no major diseases ,chronic diseases and family history.
* for children with good nutritional status: healthy,-1 <BMI z score <1; have not been treated for thyroid disease; have not used amiodarone and other drugs (including iodine supplements) during the investigation; have no major diseases ,chronic diseases and family history;

Exclusion Criteria:

long-term low-protein; long-term low-heat energy malnutrition

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 3-6 years old pre-school children are the research subjects. They were recruited in Tianjin and Shandong.
Sampling Method: Probability Sample
Enrollment: 2650 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
urinary iodine concentration | 2 weeks
  μg/L
diet iodine intake | 2 weeks
  μg/day
urinary iodine excretion | 2 weeks
  μg/day
thyroglobulin antibody | 2 weeks
  IU/mL
salt iodine concentration | 2 weeks
  μg/L
water iodine intake | 2 weeks
  μg/day
thyroid volume | 2 weeks
  ml

CONTACTS AND LOCATIONS:
Overall Officials: xiao ming Wang, Study Chair — Shandong Institute for Endemic Disease Control and Research; dong An, Study Chair — Tianjin Children's Hospital; fang Fang, Study Chair — Tianjin Medical University; na Sai, Study Chair — Tianjin Medical University
Locations (1):
- Shandong Institute for Endemic Disease Control and Research, Yuncheng, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laurberg P, Cerqueira C, Ovesen L, Rasmussen LB, Perrild H, Andersen S, Pedersen IB, Carle A. Iodine intake as a determinant of thyroid disorders in populations. Best Pract Res Clin Endocrinol Metab. 2010 Feb;24(1):13-27. doi: 10.1016/j.beem.2009.08.013. PMID 20172467
- [Background] Zimmermann MB, Boelaert K. Iodine deficiency and thyroid disorders. Lancet Diabetes Endocrinol. 2015 Apr;3(4):286-95. doi: 10.1016/S2213-8587(14)70225-6. Epub 2015 Jan 13. PMID 25591468
- [Background] Li Y, Teng D, Ba J, Chen B, Du J, He L, Lai X, Teng X, Shi X, Li Y, Chi H, Liao E, Liu C, Liu L, Qin G, Qin Y, Quan H, Shi B, Sun H, Tang X, Tong N, Wang G, Zhang JA, Wang Y, Xue Y, Yan L, Yang J, Yang L, Yao Y, Ye Z, Zhang Q, Zhang L, Zhu J, Zhu M, Ning G, Mu Y, Zhao J, Shan Z, Teng W. Efficacy and Safety of Long-Term Universal Salt Iodization on Thyroid Disorders: Epidemiological Evidence from 31 Provinces of Mainland China. Thyroid. 2020 Apr;30(4):568-579. doi: 10.1089/thy.2019.0067. Epub 2020 Mar 24. PMID 32075540
- [Background] Sang Z, Chen W, Shen J, Tan L, Zhao N, Liu H, Wen S, Wei W, Zhang G, Zhang W. Long-term exposure to excessive iodine from water is associated with thyroid dysfunction in children. J Nutr. 2013 Dec;143(12):2038-43. doi: 10.3945/jn.113.179135. Epub 2013 Oct 9. PMID 24108132
- [Background] Lee SY, Pearce EN. Reproductive endocrinology: Iodine intake in pregnancy--even a little excess is too much. Nat Rev Endocrinol. 2015 May;11(5):260-1. doi: 10.1038/nrendo.2015.28. Epub 2015 Feb 24. PMID 25707780
- [Background] Bougma K, Aboud FE, Harding KB, Marquis GS. Iodine and mental development of children 5 years old and under: a systematic review and meta-analysis. Nutrients. 2013 Apr 22;5(4):1384-416. doi: 10.3390/nu5041384. PMID 23609774
- [Background] Pearce EN, Lazarus JH, Moreno-Reyes R, Zimmermann MB. Consequences of iodine deficiency and excess in pregnant women: an overview of current knowns and unknowns. Am J Clin Nutr. 2016 Sep;104 Suppl 3(Suppl 3):918S-23S. doi: 10.3945/ajcn.115.110429. Epub 2016 Aug 17. PMID 27534632
- [Background] Zimmermann MB, Jooste PL, Mabapa NS, Mbhenyane X, Schoeman S, Biebinger R, Chaouki N, Bozo M, Grimci L, Bridson J. Treatment of iodine deficiency in school-age children increases insulin-like growth factor (IGF)-I and IGF binding protein-3 concentrations and improves somatic growth. J Clin Endocrinol Metab. 2007 Feb;92(2):437-42. doi: 10.1210/jc.2006-1901. Epub 2006 Nov 21. PMID 17118996
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Harika R, Faber M, Samuel F, Mulugeta A, Kimiywe J, Eilander A. Are Low Intakes and Deficiencies in Iron, Vitamin A, Zinc, and Iodine of Public Health Concern in Ethiopian, Kenyan, Nigerian, and South African Children and Adolescents? Food Nutr Bull. 2017 Sep;38(3):405-427. doi: 10.1177/0379572117715818. Epub 2017 Jul 6. PMID 28682645
- [Background] Lee J, Kim JH, Lee SY, Lee JH. Iodine status in Korean preschool children as determined by urinary iodine excretion. Eur J Nutr. 2014;53(2):683-8. doi: 10.1007/s00394-013-0558-y. Epub 2013 Jul 24. PMID 23881585
- [Background] Nakatsuka H, Watanabe T, Shimbo S, Sawatari H, Izumi K, Yaginuma-Sakurai K, Ikeda M. High iodine intake by preschool children in Miyagi prefecture, Japan. Environ Health Prev Med. 2014 Sep;19(5):330-8. doi: 10.1007/s12199-014-0394-6. Epub 2014 Jun 28. PMID 24972786
- [Background] Wang Y, Cui Y, Chen C, Duan Y, Wu Y, Li W, Zhang D, Li F, Hou C. Stopping the supply of iodized salt alone is not enough to make iodine nutrition suitable for children in higher water iodine areas: A cross-sectional study in northern China. Ecotoxicol Environ Saf. 2020 Jan 30;188:109930. doi: 10.1016/j.ecoenv.2019.109930. Epub 2019 Nov 11. PMID 31727496
- [Background] Chen W, Li X, Wu Y, Bian J, Shen J, Jiang W, Tan L, Wang X, Wang W, Pearce EN, Zimmermann MB, Carriquiry AL, Zhang W. Associations between iodine intake, thyroid volume, and goiter rate in school-aged Chinese children from areas with high iodine drinking water concentrations. Am J Clin Nutr. 2017 Jan;105(1):228-233. doi: 10.3945/ajcn.116.139725. Epub 2016 Dec 7. PMID 27927635
- [Background] Malvaux P, Beckers C, De Visscher M. Iodine balance studies in nongoitrous children and in adolescents on low iodine intake. J Clin Endocrinol Metab. 1969 Jan;29(1):79-84. doi: 10.1210/jcem-29-1-79. No abstract available. PMID 5762324
- [Background] Dold S, Zimmermann MB, Baumgartner J, Davaz T, Galetti V, Braegger C, Andersson M. A dose-response crossover iodine balance study to determine iodine requirements in early infancy. Am J Clin Nutr. 2016 Sep;104(3):620-8. doi: 10.3945/ajcn.116.134049. Epub 2016 Jul 27. PMID 27465383
- [Background] Tan L, Tian X, Wang W, Guo X, Sang Z, Li X, Zhang P, Sun Y, Tang C, Xu Z, Shen J, Zhang W. Exploration of the appropriate recommended nutrient intake of iodine in healthy Chinese women: an iodine balance experiment. Br J Nutr. 2019 Mar 14;121(5):519-528. doi: 10.1017/S0007114518003653. Epub 2018 Dec 11. PMID 30526700
- [Background] Yang L, Wang J, Yang J, Zhang H, Liu X, Mao D, Lu J, Gu Y, Li X, Wang H, Xu J, Tan H, Zhang H, Yu W, Tao X, Fan Y, Cai Q, Liu X, Yang X. An iodine balance study to explore the recommended nutrient intake of iodine in Chinese young adults. Br J Nutr. 2020 Dec 14;124(11):1156-1165. doi: 10.1017/S0007114520002196. Epub 2020 Jun 22. PMID 32624007
- [Background] RIGGS DS. Quantitative aspects of iodine metabolism in man. Pharmacol Rev. 1952 Sep;4(3):284-370. No abstract available. PMID 12993583
- [Background] Paul T, Meyers B, Witorsch RJ, Pino S, Chipkin S, Ingbar SH, Braverman LE. The effect of small increases in dietary iodine on thyroid function in euthyroid subjects. Metabolism. 1988 Feb;37(2):121-4. doi: 10.1016/s0026-0495(98)90004-x. PMID 3340004
- [Background] Gardner DF, Centor RM, Utiger RD. Effects of low dose oral iodide supplementation on thyroid function in normal men. Clin Endocrinol (Oxf). 1988 Mar;28(3):283-8. doi: 10.1111/j.1365-2265.1988.tb01214.x. PMID 3139337
- [Background] Sang Z, Wang PP, Yao Z, Shen J, Halfyard B, Tan L, Zhao N, Wu Y, Gao S, Tan J, Liu J, Chen Z, Zhang W. Exploration of the safe upper level of iodine intake in euthyroid Chinese adults: a randomized double-blind trial. Am J Clin Nutr. 2012 Feb;95(2):367-73. doi: 10.3945/ajcn.111.028001. Epub 2011 Dec 28. PMID 22205314
- [Background] Chen W, Zhang Y, Hao Y, Wang W, Tan L, Bian J, Pearce EN, Zimmermann MB, Shen J, Zhang W. Adverse effects on thyroid of Chinese children exposed to long-term iodine excess: optimal and safe Tolerable Upper Intake Levels of iodine for 7- to 14-y-old children. Am J Clin Nutr. 2018 May 1;107(5):780-788. doi: 10.1093/ajcn/nqy011. PMID 29722836
- [Background] Xu T, Ren Z, Li S, Tan L, Zhang W. The relationship of different levels of high iodine and goiter in school children: a meta-analysis. Nutr Metab (Lond). 2021 May 3;18(1):46. doi: 10.1186/s12986-021-00563-2. PMID 33941207
- [Background] DU Y, Gao YH, Feng ZY, Meng FG, Fan LJ, Sun DJ. Serum Thyroglobulin-A Sensitive Biomarker of Iodine Nutrition Status and Affected by Thyroid Abnormalities and Disease in Adult Populations. Biomed Environ Sci. 2017 Jul;30(7):508-516. doi: 10.3967/bes2017.067. PMID 28756810
- [Background] Andersen S, Noahsen P, Westergaard L, Laurberg P. Reliability of thyroglobulin in serum compared with urinary iodine when assessing individual and population iodine nutrition status. Br J Nutr. 2017 Feb;117(3):441-449. doi: 10.1017/S0007114517000162. Epub 2017 Feb 22. PMID 28222819
- [Background] Farebrother J, Zimmermann MB, Assey V, Castro MC, Cherkaoui M, Fingerhut R, Jia Q, Jukic T, Makokha A, San Luis TO, Wegmuller R, Andersson M. Thyroglobulin Is Markedly Elevated in 6- to 24-Month-Old Infants at Both Low and High Iodine Intakes and Suggests a Narrow Optimal Iodine Intake Range. Thyroid. 2019 Feb;29(2):268-277. doi: 10.1089/thy.2018.0321. PMID 30648484
- [Background] Stinca S, Andersson M, Erhardt J, Zimmermann MB. Development and Validation of a New Low-Cost Enzyme-Linked Immunoassay for Serum and Dried Blood Spot Thyroglobulin. Thyroid. 2015 Dec;25(12):1297-305. doi: 10.1089/thy.2015.0428. Epub 2015 Dec 1. PMID 26528830
- [Background] Chen W, Zhang Q, Wu Y, Wang W, Wang X, Pearce EN, Tan L, Shen J, Zhang W. Shift of Reference Values for Thyroid Volume by Ultrasound in 8- to 13-Year-Olds with Sufficient Iodine Intake in China. Thyroid. 2019 Mar;29(3):405-411. doi: 10.1089/thy.2018.0412. PMID 30696370